CLINICAL TRIAL: NCT06410898
Title: Assessment of Hypoxia Inducible Factor and Autophagy Related Genes in Patients With Non-Segmental Vitiligo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Rania Hassan Metwaly, Resident Dermatologist in Akhmim hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Soh-Med-24-04-014MS
Record Dates: First submitted 2024-05-02; First posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- skin biopsy from vitiligo lesion in vitiligo patient (Active Comparator): punch biopsy 5mm from vitiligo patch in vitiligo patient
  Interventions: Device: Punch Biopsy 5mm
- skin biopsy from normal skin in vitiligo patient (Active Comparator): punch biopsy 5mm from normal skin patch in vitiligo patient
  Interventions: Device: Punch Biopsy 5mm
- skin biopsy from normal skin in normal person (Active Comparator): punch biopsy 5mm from normal skin patch in normal person
  Interventions: Device: Punch Biopsy 5mm

INTERVENTIONS:
Device: Punch Biopsy 5mm — Disinfect the skin, inject local anesthesia ,insert the punch and extract the biopsy

SUMMARY:
The present study will aim to evaluate:

1. The presence of Hypoxia Inducible Factor in vitiligo patient
2. Defect of Autophagy Related Genes in vitiligo patient
3. The cross relation between Autophagy Related Genes and Hypoxia Inducible Factor in the pathogenesis of vitiligo among Egyptian patients in Sohag Governorate

ELIGIBILITY:
Inclusion Criteria:

* Adult >18 years
* With non segmental vitiligo
* A group of participants will be included as a control group

Exclusion Criteria:

* Pregnancy
* Patient with chronic inflammatory skin disorders
* patient on anti-oxidant or anti-inflammatory drugs
* patient on topical or systemic treatment for vitiligo in last 4 weeks
* patients with other autoimmune diseases
* patients with diabetes mellitus

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2024-07-25 (Estimated); Study Completion 2024-07-25 (Estimated)

PRIMARY OUTCOMES:
Assessment of Autophagy Related genes in Vitiligo patients | 2 months
  Assess Autophagy Related genes levels in skin biopsy of vitiligo patient
Assessment of Hypoxia Inducible Factor in Vitiligo patients | 2 months
  Assess level of Hypoxia Inducible factor in skin biopsy of vitiligo patient

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University hospitals, Sohag, Egypt

REFERENCES:
- [Background] Agarwal S, Ganesh S. Perinuclear mitochondrial clustering, increased ROS levels, and HIF1 are required for the activation of HSF1 by heat stress. J Cell Sci. 2020 Jul 9;133(13):jcs245589. doi: 10.1242/jcs.245589. PMID 32503939
- [Background] Artika IM, Dewi YP, Nainggolan IM, Siregar JE, Antonjaya U. Real-Time Polymerase Chain Reaction: Current Techniques, Applications, and Role in COVID-19 Diagnosis. Genes (Basel). 2022 Dec 16;13(12):2387. doi: 10.3390/genes13122387. PMID 36553654
- [Background] Bastonini E, Kovacs D, Raffa S, Delle Macchie M, Pacifico A, Iacovelli P, Torrisi MR, Picardo M. A protective role for autophagy in vitiligo. Cell Death Dis. 2021 Mar 25;12(4):318. doi: 10.1038/s41419-021-03592-0. PMID 33767135
- [Background] Ezzedine K, Lim HW, Suzuki T, Katayama I, Hamzavi I, Lan CC, Goh BK, Anbar T, Silva de Castro C, Lee AY, Parsad D, van Geel N, Le Poole IC, Oiso N, Benzekri L, Spritz R, Gauthier Y, Hann SK, Picardo M, Taieb A; Vitiligo Global Issue Consensus Conference Panelists. Revised classification/nomenclature of vitiligo and related issues: the Vitiligo Global Issues Consensus Conference. Pigment Cell Melanoma Res. 2012 May;25(3):E1-13. doi: 10.1111/j.1755-148X.2012.00997.x. PMID 22417114